CLINICAL TRIAL: NCT03159741
Title: Investigation of GLP-2 Mechanism of Action (GA-8)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirsa Skov-Jeppesen, Investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GA-8-2017
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inhibitor + GLP-2 (Experimental)
  Interventions: Other: Inhibitor + GLP-2
- Placebo + GLP-2 (Experimental)
  Interventions: Other: Placebo + GLP-2
- Placebo + GIP (Active Comparator)
  Interventions: Other: Placebo + GIP
- Placebo + Saline (Placebo Comparator)
  Interventions: Other: Placebo + Saline

INTERVENTIONS:
Other: Inhibitor + GLP-2 — Inhibitor and GLP-2 are used as study tools.
  Arms: Inhibitor + GLP-2
Other: Placebo + GLP-2 — Placebo and GLP-2 are used as study tools.
  Arms: Placebo + GLP-2
Other: Placebo + GIP — Placebo and GIP are used as study tools.
  Arms: Placebo + GIP
Other: Placebo + Saline — Placebo
  Arms: Placebo + Saline

SUMMARY:
Glucagon-like peptide-2 (GLP-2) is a naturally occuring hormone secreted to the circulation in response to food ingestion. Previous studies have shown that GLP-2 and incretins inhibit the bone resorption. However, the mechanism is unknown. In the present study we will investigate the mechanism of action using a receptor specific inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, 20 to 40 years old, caucasian, BMI 18,5 to 24,9 kg/m2

Exclusion Criteria:

* Chronic disease, smoking, medication, weight change more than 3 kg whitin the last 3 months, overweight surgery, intestinal surgery, Hgb<8,0 mmol/L, decreased renal function.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
C-terminal telopeptide (CTX) | -30 to 240 min.
  Marker of bone resorption

SECONDARY OUTCOMES:
N-terminal propeptide of type 1 procollagen (P1NP) | -30 to 240 min.
  Marker of bone formation
Osteocalcin (OC) | -30 to 240 min.
  Bone marker
Parathyroid hormone (PTH) | -30 to 240 min.
  Bone marker
Osteoprotegerin (OPG) | -30 to 240 min.
  Bone marker
Glucose-dependent insulinotropic polypeptide (GIP) | -30 to 240 min.
  GIP total and intact
Glukagon-like peptide-1 (GLP-1) and glukagon-like peptide-2 (GLP-2) | -30 to 240 min.
Glukagon and pancreatic polypeptide (PP) | -30 to 240 min.
Glucose | -30 to 240 min.
Insulin/c-pep. | -30 to 240 min.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Rosenkilde, MD, Study Director — University of Copenhagen; Sten Madsbad, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Skov-Jeppesen K, Svane MS, Martinussen C, Gabe MBN, Gasbjerg LS, Veedfald S, Bojsen-Moller KN, Madsbad S, Holst JJ, Rosenkilde MM, Hartmann B. GLP-2 and GIP exert separate effects on bone turnover: A randomized, placebo-controlled, crossover study in healthy young men. Bone. 2019 Aug;125:178-185. doi: 10.1016/j.bone.2019.05.014. Epub 2019 May 15. PMID 31100534